CLINICAL TRIAL: NCT01046760
Title: Scholar Performance and Praxis Assessment in Children With Rolandic Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Ecila Paula dos Mesquita de Oliveira, UNICAMP
Other Study IDs: 21 CFR 50.3.
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-10

CONDITIONS: Rolandic Epilepsy; Apraxia
Keywords: epilepsy; language; childhood; praxis
MeSH Terms: conditions — Epilepsy, Rolandic; Apraxias; Epilepsy; Language

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Rolandic Epilepsy: Patients older than seven years old with clinical and electroencephalographic diagnosis of Rolandic Epilepsy
  Interventions: Behavioral: Language Assessment

INTERVENTIONS:
Behavioral: Language Assessment — Patients underwent an assessment performed with School Performance Test, Syntactic Awareness Test and a Peabody Picture Vocabulary Test.
  Other Names: Children with epilepsy, language impairment and dyslexia

SUMMARY:
Rolandic Epilepsy is the most common form of childhood epilepsy. It is classified as idiopathic, age-related epilepsy syndrome with benign evolution. The absence of neuropsychological impairment is part of the criteria of benignity of this epilepsy syndrome. However recently have been suggested several deficits related to attention and language. The purpose of this study was assess school performance and to investigate problems of praxis in patients with rolandic epilepsy as compared to a control group composed of normal children with age, gender and educational level equivalents.

DETAILED DESCRIPTION:
Method: Nineteen patients aged between 7 and 12 years underwent clinical neurological evaluation, psychological assessment, through Weschsler Scales of Intelligence and language evaluation, to assess the academic performance and research of the presence or absence of praxis difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rolandic epilepsy using clinical, EEG and neuroimaging findings
* Patients had neurological, ophthalmic and auditory unchanged, and intelligence quotient (IQ) equal to or above 80.
* All parents signed the consent form, authorizing the participation of their children (as) in the search.

Exclusion Criteria:

* With oral language and writing of the following tables, whereas the DSM-IV: pervasive developmental disorders, cerebral palsy child acquired aphasia, hearing impairment (including mild conductive hearing loss), progressive disease
* What not signed the consent form.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Amongst patients with rolandic epilepsy assisted at the Clinic of Neurological-Psychological-Language in childhood of Hospital de Clínicas of Universidade Estadual de Campinas (Unicamp).
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Our data will indicate the group performance in tests of writing, arithmetic and reading. | one year

SECONDARY OUTCOMES:
Another important aspect was the absence of orofacial apraxia in children with epilepsy. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Marilisa Guerreiro, doctor, Study Chair — University of Campinas, Brazil
Locations (1):
- Clinical Hospital, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Oliveira EP, Neri ML, Medeiros LL, Guimaraes CA, Guerreiro MM. School performance and praxis assessment in children with Rolandic Epilepsy. Pro Fono. 2010 Jul-Sep;22(3):209-14. doi: 10.1590/s0104-56872010000300009. English, Portuguese. PMID 21103707
- See also: CARACTERIZACAO DAS MANIFESTACOES NEUROPSICOLINGUISTICAS EM CRIANCAS COM EPILEPSIA ROLANDICA. — http://internet.aquila.fapesp.br/agilis/